CLINICAL TRIAL: NCT03477955
Title: PEEK Versus Silicon Interspinous Spacer for Reduction of Supradjacent Segment Degeneration Following Decompression and Short-Segment Instrumentation for Degenerative Lumbar Spinal Stenosis
Brief Title: PEEK Versus Silicon Interspinous Spacer for Reduction of Supradjacent Segment Degeneration
Acronym: WallisvsDiam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Collaborators: St. Andrew's General Hospital, Patras, Greece (Other)
Responsible Party: Principal Investigator, Vasileios Syrimpeis, Orthopaedic Surgeon, University Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WALLIS2018
Record Dates: First submitted 2018-03-03; First posted 2018-03-27 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Adjacent Segment Degeneration
Keywords: spinopelvic alignment; short lumbosacral instrumentation; PEEK; silicon spacer

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peek Group (Active Comparator): Patients that received PEEK interspinous spacer
  Interventions: Procedure: PEEK interspinous spacer
- Silicon Group (Active Comparator): Patients that received Silicon interspinous spacer and did not receive PEEK interspinous spacer
  Interventions: Procedure: PEEK interspinous spacer
- Control Group (Active Comparator): Patients that did not receive PEEK interspinous spacer nor Silicon interspinous spacer
  Interventions: Procedure: PEEK interspinous spacer

INTERVENTIONS:
Procedure: PEEK interspinous spacer — To study the Adjacent Segment Degeneration incidence in the supradjacent segment following short lumbar fusion between PEEK and Silicon Interspinous spacers.
  Other Names: Silicon interspinous spacer

SUMMARY:
A retrospective study that aims to report Adjacent Segment Degeneration (ASD) incidence and spinopelvic balance in short lumbosacral instrumentation for degenerative lumbar spinal stenosis. Although ASD is a common complication following lumbar fusion, the effect of an Interspinous Spacer (IS) in the supradjacent segment in short lumbosacral instrumented fusion and its interaction with spinopelvic balance has not been studied adequately.

DETAILED DESCRIPTION:
Methods From 55 consecutive age-, diagnosis- and gender- matched patients aged 60±11 years, 17 (Group R) received PEEK IS; 18 (Group S) received Silicon IS and compared with 20 controls (Group C) without receiving any IS. The functional outcome was evaluated with VAS and ODI. Spinopelvic balance was evaluated using SVA, T12-S1 LL, SS, PT, PI and supradjacent segment disc heights. All spines were preoperatively balanced.

ELIGIBILITY:
Inclusion Criteria:

Preoperative MRI with degeneration grades<III at the 1st supradjacent lumbar segment.

Exclusion Criteria:

* Body mass index≥40kg/m*m
* Severe osteoporosis
* Lumbar fracture
* Preoperative SVA>4cm
* Spondylolisthesis grades>II or spondylolytic lesion and acquired spinous process insufficiency in the supradjacent segment cephalad to instrumentation

Ages: 49 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2006-04 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Quality of Life | Three years
  Oswestry Disability Index scale (0-100)

SECONDARY OUTCOMES:
Disc heights | Three years
  Measured in cm
Sacral Slope | Three years
  Measured in degrees
Pain | Three years
  Visual Analog Scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Korovessis, PhD, Principal Investigator — General Hospital of Patras

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Korovessis P, Syrimpeis V, Tsekouras V, Vardakastanis K, Fennema P. PEEK versus Silicon Interspinous Spacer for Reduction of Supradjacent Segment Degeneration following Decompression and Short-Segment Instrumentation for Degenerative Lumbar Spinal Stenosis. Adv Orthop. 2018 Aug 8;2018:1623647. doi: 10.1155/2018/1623647. eCollection 2018. PMID 30174959